CLINICAL TRIAL: NCT07243145
Title: Analysis of the Impact of Contemporary Subgingival Debridement Techniques on Immunological Biomarkers in Gingival Crevicular Fluid
Status: Completed | Type: Observational
Sponsor: Selcen Ozcan Bulut (Other)
Collaborators: Nigde Omer Halisdemir University (Other); Niğde Ömer Halisdemir University (Unknown)
Responsible Party: Sponsor-Investigator, Selcen Ozcan Bulut, Nigde Omer Halisdemir University, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: 2023/87
Record Dates: First submitted 2025-05-29; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Peridontal Disease; Periodontal Inflammation; Periodontitis, Adult
Keywords: periodontitis; guided biofilm therapy; non surgical periodontal treatment; Gingival Crevicular Fluid
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1.Group: The Conventional Treatment: Cavitron and Gracey curette (the standard technique) was utilized for subgingival debridement
- 2. group: Guided biofilm therapy: Subgingival debridement was carried out using the GBT approach, which involved following the protocol's directions properly.

SUMMARY:
AIM: This prospective clinical study aimed to evaluate the efficacy of two distinct non-surgical periodontal therapy modalities in patients diagnosed with Stage 1 and Stage 2 periodontitis.

METHOD: The study comprised 80 nonsmoking, systemically healthy volunteers. Patients were divided into two groups at random: the Guided Biofilm Therapy (GBT) group and the convetional therapy group, which included Gracey curette and an ultrasonic device. All patients were assessed before and one and three months after therapy for clinical characteristics like pocket depth, Gingival Index (GI), Plaque Index (PI), Bleeding on Probing Index (BOP), and the levels of IL-1β, IL-10, TNF-α, and MMP-8 in gingival crevicular fluid (GCF).

RESULTS: ... CONCLUSION:...

DETAILED DESCRIPTION:
AIM: This prospective clinical study aimed to evaluate the efficacy of two distinct non-surgical periodontal therapy modalities in patients diagnosed with Stage 1 and Stage 2 periodontitis.

METHOD: The study comprised 80 nonsmoking, systemically healthy volunteers. Patients were divided into two groups at random: the Guided Biofilm Therapy (GBT) group and the convetional therapy group, which included Gracey curette and an ultrasonic device. All patients were assessed before and one and three months after therapy for clinical characteristics like pocket depth, Gingival Index (GI), Plaque Index (PI), Bleeding on Probing Index (BOP), and the levels of IL-1β, IL-10, TNF-α, and MMP-8 in gingival crevicular fluid (GCF).

RESULTS: ... CONCLUSION:...

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (no known chronic diseases)
* Completed periodontal diagnostic data (Gingival Index, Plaque Index, Periodontal pocket depths, Attachment loss, Radiological data, and Bone loss data)
* Did not take anti-inflammatory drugs in the previous month
* Volunteered to participate with Stage 1-2 periodontitis.

Exclusion Criteria:

* Patients with systemic diseases
* Pregnant or lactating patients
* Smokers
* Patients who did not wish to participate in the study were excluded

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who applied to Niğde Ömer Halisdemir University Faculty of Dentistry Periodontics Clinic between 15.10.2024 and 15.12.2024 for periodontal treatment, volunteered to participate in the study and met the following criteria were included in the study. Written consent was obtained from volunteer patients for the research.
  The patients were evaluated by a single periodontologist (SND), and patients with mild to moderate periodontitis (Stage 1-2) who required supragingival and subgingival calculus removal were included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Gingival index | baseline
  All teeth are evaluated on 4 surfaces (distal, buccal, mesial, lingual) and the average is calculated.
  0= Normal gingiva
  1. Mild inflammation - minor color change, minor edema. No bleeding after probing.
  2. Moderate inflammation - redness, edema and shine. Bleeding after probing.
  3. Severe inflammation - significant redness and edema. Ulceration. Spontaneous bleeding tendency.
Gingival index | 1st month
  All teeth are evaluated on 4 surfaces (distal, buccal, mesial, lingual) and the average is calculated.
  0= Normal gingiva
  1. Mild inflammation - minor color change, minor edema. No bleeding after probing.
  2. Moderate inflammation - redness, edema and shine. Bleeding after probing.
  3. Severe inflammation - significant redness and edema. Ulceration. Spontaneous bleeding tendency.
Gingival index | 3rd month
  All teeth are evaluated on 4 surfaces (distal, buccal, mesial, lingual) and the average is calculated.
  0= Normal gingiva
  1. Mild inflammation - minor color change, minor edema. No bleeding after probing.
  2. Moderate inflammation - redness, edema and shine. Bleeding after probing.
  3. Severe inflammation - significant redness and edema. Ulceration. Spontaneous bleeding tendency.
IL-1β | baseline
  A single specialist physician took GCF measurements at baseline, one month, and three months from the tooth with the deepest pocket identified at baseline before treatment in patients with periodontitis. In short, the region was isolated using cotton pads, and the plaque was removed using cotton pellets. After that, 20 cm of mild air drying was applied. Strips of absorbent paper (Periopaper®, Proflow Inc., Amityville, NY, USA) were used to obtain GCF samples. The strips were positioned for 30 seconds after being carefully inserted into the gingival sulcus/periodontal pocket until a small amount of resistance was felt. Strips tainted with blood were thrown away. Before being used for laboratory testing, each subject's strips were gathered, combined, and kept at -80 °C (Ultra Low-Temperature Freezer, New Brunswick Scientific).
  As directed by the manufacturer, enzyme-linked immunosorbent assay (ELISA) kits were used to measure the levels of IL-1β, TNF-alpha, IL-10, and MMP-8 in GCF
IL-1β | 1st month
  A single specialist physician (SOB) took GCF measurements at baseline, one month, and three months from the tooth with the deepest pocket identified at baseline before treatment in patients with periodontitis. In short, the region was isolated using cotton pads, and the plaque was removed using cotton pellets. After that, 20 cm of mild air drying was applied. Strips of absorbent paper (Periopaper®, Proflow Inc., Amityville, NY, USA) were used to obtain GCF samples. The strips were positioned for 30 seconds after being carefully inserted into the gingival sulcus/periodontal pocket until a small amount of resistance was felt. Strips tainted with blood were thrown away. Before being used for laboratory testing, each subject's strips were gathered, combined, and kept at -80 °C (Ultra Low-Temperature Freezer, New Brunswick Scientific).
  As directed by the manufacturer, enzyme-linked immunosorbent assay (ELISA) kits were used to measure the levels of IL-1β, TNF-alpha, IL-10, and MMP-8 in GCF
IL-1β | 3rd month
  A single specialist physician (SOB) took GCF measurements at baseline, one month, and three months from the tooth with the deepest pocket identified at baseline before treatment in patients with periodontitis. In short, the region was isolated using cotton pads, and the plaque was removed using cotton pellets. After that, 20 cm of mild air drying was applied. Strips of absorbent paper (Periopaper®, Proflow Inc., Amityville, NY, USA) were used to obtain GCF samples. The strips were positioned for 30 seconds after being carefully inserted into the gingival sulcus/periodontal pocket until a small amount of resistance was felt. Strips tainted with blood were thrown away. Before being used for laboratory testing, each subject's strips were gathered, combined, and kept at -80 °C (Ultra Low-Temperature Freezer, New Brunswick Scientific).
  As directed by the manufacturer, enzyme-linked immunosorbent assay (ELISA) kits were used to measure the levels of IL-1β, TNF-alpha, IL-10, and MMP-8 in GCF

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)